CLINICAL TRIAL: NCT02320877
Title: Evaluation of the Overall Effectiveness Including Cardiovascular Effects of the Custom-made, Titratable Duoblock Flex SomnoDent® MAS in the Treatment of Obstructive Sleep Apnea
Brief Title: Evaluation of the Cardiovascular Effects of the MAS in the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Ethisch Comité UZ Antwerpen, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B300201422483
Record Dates: First submitted 2014-11-24; First posted 2014-12-19 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: OSA
MeSH Terms: interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mandibular Advancement Device (Experimental): Mandibular advancement Devices are worn intra-orally at night in order to advance the mandible and to reduce the collapsibility of the upper airway.
  Interventions: Device: Mandibular Advancement Device (Somnomed Flex)

INTERVENTIONS:
Device: Mandibular Advancement Device (Somnomed Flex) — The SomnoDent Flex™ MAS is a custom-made, titratable MAS that is validated in randomized controlled trials described in literature
  Other Names: Somnomed Flex

SUMMARY:
In this prospective trial 50 patients, diagnosed with moderate to severe obstructive sleep apnea (OSA) (AHI > 15/h sleep) will be included and treated with mandibular advancement devices (MAD). These patients will undergo cardiovascular examination; echocardiography and 24h-blood pressure monitoring, on top of the normal clinical evaluation of OSA patients. These cardiovascular examinations will take place before and during MAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 15 events/hour
* No other active OSA therapy in the 3 months preceding inclusion
* Willing to participate after informed consent
* Positive advice on OAT after DISE

Exclusion Criteria:

* Insufficient teeth to support the device
* Periodontal problems including tooth mobility
* Active temporomandibular joint dysfunction
* Limited maximum protrusive capacity (< 6 mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
cardiovascular outcome - interventricular septum thickness | 1 year
  interventricular septum thickness
cardiovascular outcome - ventricular dilatation | 1 year
  ventricular dilatation
cardiovascular outcome - cardiac strain | 1 year
  cardiac strain. This will be measured on speckle tracking echocardiopgraphy (STE). STE is an echocardiographic imaging technique that analyzes the motion of heart tissue by using ultrasound waves to generate interference patterns and natural acoustic reflections. These reflections, also described as ''speckles'', are tracked consecutively frame to frame and ultimately resolved into angle-independent two-dimensional and three-dimensional strain-based sequences (3D). These sequences provide both quantitative and qualitative information regarding heart tissue deformation and motion.
cardiovascular outcome - stroke volume | 1 year
  stroke volume

SECONDARY OUTCOMES:
OSA efficacy: apnea-hypopnea index | 1 year
  benefit in apnea-hypopnea index
Therapy compliance | 1 year
  Therapy compliance will be objectively monitored12 using 2 microsensors (Dentitrac®, Braebon Medical Corporation, Kanata, Ontario, Canada; TheraMon, IFT Handels- und Entwicklungsgesellschaft GmbH, Handelsagentur Gschladt, Hargelsberg, Austria) embedded in the OAm as well as by self-reporting
efficacy on subjective complaints: epworth sleepiness scale | 1 year
  daytime sleepiness measured using epworth sleepiness scale
efficacy on subjective complaints: visual analogue scale for snoring | 1 year
  visual analogue scale for snoring

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Dieltjens M, Vanderveken OM, Shivalkar B, Van Haesendonck G, Kastoer C, Heidbuchel H, Braem MJ, Van De Heyning CM. Mandibular advancement device treatment and reverse left ventricular hypertrophic remodeling in patients with obstructive sleep apnea. J Clin Sleep Med. 2022 Mar 1;18(3):903-909. doi: 10.5664/jcsm.9766. PMID 34728052